CLINICAL TRIAL: NCT01018134
Title: A Double-Blind, Vehicle-Controlled, Randomized, Dose Ranging, Multiple-Site Clinical Study to Evaluate the Efficacy and Safety of Desoximetasone Topical Sprays (0.05%, 0.25%) in Patients With Moderate to Severe Plaque Psoriasis
Brief Title: Desoximetasone Spray 0.05%, 0.25%; Dose Ranging Study
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Sun Pharmaceutical Industries, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: DSXS 0906.00; 70915004 (Other: Novum PRS)
Record Dates: First submitted 2009-11-19; First posted 2009-11-23 (Estimated); Results first posted 2014-08-05 (Estimated); Last update posted 2014-08-05 (Estimated); Status verified 2014-07

CONDITIONS: Psoriasis
Keywords: Psoriasis; Topical corticosteroids; Plaque psoriasis
MeSH Terms: conditions — Psoriasis | interventions — Desoximetasone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Desoximetasone 0.05% once daily (Experimental): Desoximetasone topical spray 0.05% administered once daily to affected area
  Interventions: Drug: Desoximetasone 0.05% once daily
- Desoximetasone 0.05% twice daily (Experimental): Desoximetasone topical spray 0.05% administered twice daily to affected area
  Interventions: Drug: Desoximetasone 0.05% twice daily
- Desoximetasone 0.25% once daily (Experimental): Desoximetasone topical spray 0.25% administered once daily to affected area
  Interventions: Drug: Desoximetasone 0.25% once daily
- Desoximetasone 0.25% twice daily (Experimental): Desoximetasone topical spray 0.25% administered twice daily to affected area
  Interventions: Drug: Desoximetasone 0.25% once daily
- Vehicle once daily (Placebo Comparator): Vehicle administered to affected areas once daily
  Interventions: Drug: Vehicle once daily
- Vehicle twice daily (Placebo Comparator): Vehicle administered to affected areas twice daily
  Interventions: Drug: Vehicle twice daily

INTERVENTIONS:
Drug: Desoximetasone 0.05% once daily — Desoximetasone topical spray 0.05% administered to affected area once daily for 28 days
  Arms: Desoximetasone 0.05% once daily
Drug: Desoximetasone 0.05% twice daily — Desoximetasone topical spray 0.05% administered to affected area twice daily for 28 days
  Arms: Desoximetasone 0.05% twice daily
Drug: Desoximetasone 0.25% once daily — Desoximetasone topical spray 0.25% administered to affected area once daily for 28 days
  Arms: Desoximetasone 0.25% once daily
Drug: Desoximetasone 0.25% once daily — Desoximetasone topical spray 0.25% administered to affected areas twice daily for 28 days
  Arms: Desoximetasone 0.25% twice daily
Drug: Vehicle once daily — Vehicle topical spray administered to affected areas once daily for 28 days
  Arms: Vehicle once daily
Drug: Vehicle twice daily — Vehicle topical spray administered to affected areas twice daily for 28 days
  Arms: Vehicle twice daily

SUMMARY:
The objectives of this study are to evaluate the efficacy and safety of two dosing regimens of desoximetasone 0.05% and 0.25% topical sprays as compared to a vehicle spray in patients with moderate to severe plaque psoriasis.

ELIGIBILITY:
Inclusion Criteria:

* Have a definite clinical diagnosis of stable plaque psoriasis involving ≥ 10% of the body surface area (BSA).
* Have a combined total lesion severity score (TLSS) of ≥ 7 for the target lesion.
* Have a plaque elevation score ≥ 3 of (moderate) for the target lesion.
* The target lesion must have an area of at least 5 cm².
* Have a Physicians Global Assessment (PGA) score of 3 (moderate) or 4 (severe) at baseline for the overall disease severity.

Exclusion Criteria:

* Pregnancy
* Current diagnosis of other types of psoriasis other than stable plaque psoriasis or has psoriasis of any kind of the face or scalp that will require active treatment during the study.
* History of psoriasis that has been unresponsive to topical corticosteroid therapy.
* Dermatological conditions that may interfere with the clinical assessments of the signs and symptoms of psoriasis.
* Allergy or sensitivity to corticosteroids or history of any drug hypersensitivity or intolerance which would compromise the safety of the patient or the results of the study.
* Any condition that would place the study patient at undue risk by participation in the study.
* Radiation therapy, antineoplastic agents or immunosuppressant medication within 4 weeks prior to the first dose of study drug.
* Treatment with any systemic or photo antipsoriatic therapy, within 8 weeks of the first dose of study drug.
* Treatment within 12 weeks (or five half lives, whichever is less) prior to the first dose of study drug with any biological therapies for psoriasis.
* Systemic steroids within 4 weeks of the first dose of the study drug. The use of inhaled or intranasal corticosteroids is acceptable as long as usage has been stable for at least 2 weeks prior to the first dose of study drug and will be continued during the study.
* Hormonal contraceptives for less than one complete cycle prior to entering the study.
* Topical antipsoriatic agents of any kind or any topical corticosteroids for any reason within 2 weeks prior to first use of study drug. Nonprescription antipsoriatic shampoos used only on the scalp will be allowed during the study.
* Receipt of any drug as part of a research study within 30 days prior to first dosing.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 151 (Actual)
Dates: Start 2009-11; Primary Completion 2010-05 (Actual); Study Completion 2010-05 (Actual)

CONTACTS AND LOCATIONS:
Locations (7):
- United States (7):
  - Investigator Site, Miami, Florida
  - Investigator Site, Martinez, Georgia
  - Investigator Site, Olathe, Kansas
  - Investigator Site, Wichita, Kansas
  - Investigator Site, Albuquerque, New Mexico
  - Investigator Site, Cincinnati, Ohio
  - Investigator Site, Simpsonville, South Carolina

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Desoximetasone 0.05% Once Daily | Desoximetasone 0.05% Twice Daily | Desoximetasone 0.25% Once Daily | Desoximetasone 0.25% Twice Daily | Vehicle Once Daily | Vehicle Twice Daily
Started | 30 | 31 | 30 | 29 (30 enrolled patients, one who did not use the study medication was excluded from all analyses) | 15 | 15
Completed | 30 | 30 | 29 | 29 | 15 | 15
Not Completed | 0 | 1 | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Desoximetasone 0.05% Once Daily | Desoximetasone 0.05% Twice Daily | Desoximetasone 0.25% Once Daily | Desoximetasone 0.25% Twice Daily | Vehicle Once Daily | Vehicle Twice Daily | Total
Number analyzed (Participants) | 30 | 31 | 30 | 29 | 15 | 15 | 150
Age, Continuous [Mean (Standard Deviation); unit: years] | 53.60 (15.21) | 45.06 (13.04) | 51.60 (12.67) | 50.62 (14.54) | 53.53 (12.92) | 49.60 (13.30) | 50.66 (13.61)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 12 | 13 | 14 | 11 | 1 | 7 | 58
  Male | 18 | 18 | 16 | 18 | 14 | 8 | 92
Region of Enrollment [Number; unit: participants]
  United States | 30 | 31 | 30 | 29 | 15 | 15 | 150

OUTCOME MEASURES:

1. Primary Outcome: Number of Participants in Each Treatment Group With Clinical Cure: Physician's Global Assessment (PGA) Score = 0 or 1 at Day 28
Description: The primary endpoint was the proportion of patients in each treatment group who were considered a Clinical Success (PGA score of 0 or 1) at Day 28 for each of the three signs/symptoms (i.e., scaling, erythema and plaque elevation)
  The primary measure of efficacy was evaluated using those patients eligible for inclusion in the ITT population.
  On a seven point grade PGA scale a patient will be considered a Clinical Success if: the patient's PGA score is 0 or 1.
  A score of 0 = Clear or 1= Almost Clear was considered clinical success.
  A patient will be considered a Clinical Failure if: the patient's PGA score is > 1, the patient was considered to have an insufficient therapeutic response
Time Frame: 28 days
Population: The primary measure of efficacy was based on the ITT population. One hundred fifty (150) patients used the study medication and were included in the analysis of safety. Two patients withdrew consent and did not have end of study efficacy procedures performed and were excluded from the efficacy analysis.
Measure: Number; unit: percentage of participants
Arm/Group | Desoximetasone 0.05% Once Daily | Desoximetasone 0.05% Twice Daily | Desoximetasone 0.25% Once Daily | Desoximetasone 0.25% Twice Daily | Vehicle Once Daily | Vehicle Twice Daily
Number analyzed (Participants) | 30 | 30 | 29 | 29 | 15 | 15
percentage of participants | 13.33 | 10.00 | 20.69 | 37.93 | 6.67 | 6.67
Statistical Analysis 1: Comparison: Desoximetasone 0.05% Once Daily vs Vehicle Once Daily; Test type: Superiority or Other; p = 0.4261, t-test, 1 sided
Statistical Analysis 2: Comparison: Desoximetasone 0.05% Twice Daily vs Vehicle Twice Daily; Test type: Superiority or Other; p = 0.4219, t-test, 1 sided
Statistical Analysis 3: Comparison: Desoximetasone 0.25% Once Daily vs Vehicle Once Daily; Test type: Superiority or Other; p = 0.1826, t-test, 1 sided
Statistical Analysis 4: Comparison: Desoximetasone 0.25% Twice Daily vs Vehicle Twice Daily; Test type: Superiority or Other; p = 0.0090, t-test, 1 sided — Statistically significant difference between treatment groups
Statistical Analysis 5: Comparison: Desoximetasone 0.05% Once Daily vs Desoximetasone 0.25% Once Daily; Test type: Superiority or Other; p = 0.3421, t-test, 1 sided
Statistical Analysis 6: Comparison: Desoximetasone 0.05% Twice Daily vs Desoximetasone 0.25% Twice Daily; Test type: Superiority or Other; p = 0.0100, t-test, 1 sided — Statistically significant difference between treatment groups
Statistical Analysis 7: Comparison: Desoximetasone 0.05% Once Daily vs Desoximetasone 0.05% Twice Daily; Test type: Superiority or Other; p = 0.2103, t-test, 1 sided
Statistical Analysis 8: Comparison: Desoximetasone 0.25% Once Daily vs Desoximetasone 0.25% Twice Daily; Test type: Superiority or Other; p = 0.1200, t-test, 1 sided

2. Primary Outcome: Number of Participants in Each Treatment Group With Treatment Success for the Target Lesion (Total Lesion Severity Scale (TLSS) a Score of 0 or 1).
Description: The proportion of patients in each treatment group who were considered a Treatment Success for the target lesion (a score of 0 or 1 for each of the three signs/symptoms (i.e., scaling, erythema and plaque elevation)) at Day 28.
  Each component was given a score using the following scale: 0=clear, 1=Almost Clear, 2=Mild, 3=Moderate, 4=Severe, 5=Very Severe., with increasing score reflecting increased lesion severity. The TLS score is calculated as the sum of the 3 components.
  A TLS score of 0 = Clear or 1= Almost Clear was considered treatment success.
Time Frame: Day 28
Population: as for outcome 1
Measure: Number; unit: percentage of Participants
Arm/Group | Desoximetasone 0.05% Once Daily | Desoximetasone 0.05% Twice Daily | Desoximetasone 0.25% Once Daily | Desoximetasone 0.25% Twice Daily | Vehicle Once Daily | Vehicle Twice Daily
Number analyzed (Participants) | 30 | 30 | 29 | 29 | 15 | 15
percentage of Participants | 6.67 | 16.67 | 34.48 | 31.03 | 6.67 | 6.67
Statistical Analysis 1: Comparison: Desoximetasone 0.05% Once Daily vs Vehicle Once Daily; Test type: Superiority or Other; p = 0.2631, t-test, 1 sided
Statistical Analysis 2: Comparison: Desoximetasone 0.05% Twice Daily vs Vehicle Twice Daily; Test type: Superiority or Other; p = 0.2968, t-test, 1 sided
Statistical Analysis 3: Comparison: Desoximetasone 0.25% Once Daily vs Vehicle Once Daily; Test type: Superiority or Other; p = 0.0186, t-test, 1 sided — statistically significant difference between treatment groups
Statistical Analysis 4: Comparison: Desoximetasone 0.25% Twice Daily vs Vehicle Twice Daily; Test type: Superiority or Other; p = 0.0361, t-test, 1 sided — statistically significant difference between treatment groups
Statistical Analysis 5: Comparison: Desoximetasone 0.05% Once Daily vs Desoximetasone 0.25% Once Daily; Test type: Superiority or Other; p = 0.0070, t-test, 1 sided — statistically significant difference between treatment groups
Statistical Analysis 6: Comparison: Desoximetasone 0.05% Twice Daily vs Desoximetasone 0.25% Twice Daily; Test type: Superiority or Other; p = 0.1583, t-test, 1 sided
Statistical Analysis 7: Comparison: Desoximetasone 0.05% Once Daily vs Desoximetasone 0.05% Twice Daily; Test type: Superiority or Other; p = 0.2078, t-test, 1 sided
Statistical Analysis 8: Comparison: Desoximetasone 0.25% Once Daily vs Desoximetasone 0.25% Twice Daily; Test type: Superiority or Other; p = 0.2878, t-test, 1 sided

3. Secondary Outcome: Mean Change From Baseline in PGA Score at Day 28 Using the ITT
Description: Physician Global Assessment (PGA) of Psoriasis is scored based on dermatologist's assessment of disease averaged over all lesions of face, genitals, or intertriginous area (i.e., breast fold, gluteal crease, axilla). Overall lesions were graded for plaque formation, induration, erythema, and scaling; range: 0 (clear) to 5 (very severe). The severity score was summed and averaged after which the total average is rounded to the nearest whole number score to determine the PGA score and category (0=clear; 1=almost clear; 2=mild; 3=moderate; and 4=severe; 5=very severe). PGA response was defined as 0 (clear) or 1 (almost clear) Higher scores indicate greater severity of disease.
Time Frame: Day 28
Population: The Intent-to-Treat (ITT) population was used for the secondary endpoint analysis.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Desoximetasone 0.05% Once Daily | Desoximetasone 0.05% Twice Daily | Desoximetasone 0.25% Once Daily | Desoximetasone 0.25% Twice Daily | Vehicle Once Daily | Vehicle Twice Daily
Number analyzed (Participants) | 30 | 30 | 29 | 29 | 15 | 15
units on a scale | 0.63 (0.93) | 0.57 (0.68) | 0.86 (0.79) | 1.24 (0.99) | 0.40 (0.74) | 0.67 (0.62)
Statistical Analysis 1: Comparison: Desoximetasone 0.05% Once Daily vs Vehicle Once Daily; Test type: Superiority or Other; p = 0.2713, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Desoximetasone 0.05% Twice Daily vs Vehicle Twice Daily; Test type: Superiority or Other; p = 0.2689, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Desoximetasone 0.25% Once Daily vs Vehicle Once Daily; Test type: Superiority or Other; p = 0.0419, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Desoximetasone 0.25% Twice Daily vs Vehicle Twice Daily; Test type: Superiority or Other; p = 0.0309, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Desoximetasone 0.05% Once Daily vs Desoximetasone 0.25% Once Daily; Test type: Superiority or Other; p = 0.1126, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Desoximetasone 0.05% Twice Daily vs Desoximetasone 0.25% Twice Daily; Test type: Superiority or Other; p = 0.0033, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Desoximetasone 0.05% Once Daily vs Desoximetasone 0.05% Twice Daily; Test type: Superiority or Other; p = 0.4967, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Desoximetasone 0.25% Once Daily vs Desoximetasone 0.25% Twice Daily; Test type: Superiority or Other; p = 0.0749, Wilcoxon (Mann-Whitney)

4. Secondary Outcome: Mean Change From Baseline in Total Lesion Severity Score (TLSS) at Day 28
Description: Each lesion was evaluated for 3 components: erythema, plaque elevation, and scaling. Each component was given a score using the following scale: 0=clear, 1=Almost Clear, 2=Mild, 3=Moderate, 4=Severe, 5=Very Severe., with increasing score reflecting increased lesion severity. The TLS score is calculated as the sum of the 3 components.
Time Frame: Day 28
Population: The Intent-to-Treat (ITT) population was used for the secondary efficacy analysis after 28 days of treatment.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Desoximetasone 0.05% Once Daily | Desoximetasone 0.05% Twice Daily | Desoximetasone 0.25% Once Daily | Desoximetasone 0.25% Twice Daily | Vehicle Once Daily | Vehicle Twice Daily
Number analyzed (Participants) | 30 | 30 | 29 | 29 | 15 | 15
units on a scale | 2.33 (2.51) | 2.70 (2.05) | 3.79 (3.20) | 4.55 (3.03) | 2.80 (2.21) | 3.00 (1.81)
Statistical Analysis 1: Comparison: Desoximetasone 0.05% Once Daily vs Vehicle Once Daily; Test type: Superiority or Other; p = 0.2442, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Desoximetasone 0.05% Twice Daily vs Vehicle Twice Daily; Test type: Superiority or Other; p = 0.2664, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Desoximetasone 0.25% Once Daily vs Vehicle Once Daily; Test type: Superiority or Other; p = 0.1328, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Desoximetasone 0.25% Twice Daily vs Vehicle Twice Daily; Test type: Superiority or Other; p = 0.0528, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Desoximetasone 0.05% Once Daily vs Desoximetasone 0.25% Once Daily; Test type: Superiority or Other; p = 0.0297, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Desoximetasone 0.05% Twice Daily vs Desoximetasone 0.25% Twice Daily; Test type: Superiority or Other; p = 0.0093, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Desoximetasone 0.05% Once Daily vs Desoximetasone 0.05% Twice Daily; Test type: Superiority or Other; p = 0.2230, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Desoximetasone 0.25% Once Daily vs Desoximetasone 0.25% Twice Daily; Test type: Superiority or Other; p = 0.1924, Wilcoxon (Mann-Whitney)

5. Secondary Outcome: Mean Change From Baseline in %Body Surface Area (%BSA) Affected at Day 28 (or Early Termination).
Description: Body Surface Area (BSA) is a numerical score used to measure the physician's assessment of the percentage of the participant's total BSA involved with psoriasis.
  BSA = SQRT ((height (cm) X weight (kg))/3600) BSA is in m2, W is weight in kg, and H is height in cm. Total body Surface Area (BSA) in meters squared
  %Body Surface Area Affected the "Rule of Nine" was be used.
Time Frame: Day 28
Population: The Intent-to-Treat (ITT) population was used for the secondary efficacy analysis after 28 days of treatment.
Measure: Mean (Standard Deviation); unit: percentage of Body Surface Area Affected
Arm/Group | Desoximetasone 0.05% Once Daily | Desoximetasone 0.05% Twice Daily | Desoximetasone 0.25% Once Daily | Desoximetasone 0.25% Twice Daily | Vehicle Once Daily | Vehicle Twice Daily
Number analyzed (Participants) | 30 | 30 | 29 | 29 | 15 | 15
percentage of Body Surface Area Affected | 1.20 (2.44) | 0.00 (0.69) | 1.31 (2.38) | 2.76 (3.92) | 0.60 (2.06) | 0.33 (1.35)
Statistical Analysis 1: Comparison: Desoximetasone 0.05% Once Daily vs Vehicle Once Daily; Test type: Superiority or Other; p = 0.2397, Wilcoxon (Mann-Whitney)
Statistical Analysis 2: Comparison: Desoximetasone 0.05% Once Daily vs Vehicle Twice Daily; Test type: Superiority or Other; p = 0.3794, Wilcoxon (Mann-Whitney)
Statistical Analysis 3: Comparison: Desoximetasone 0.25% Once Daily vs Vehicle Once Daily; Test type: Superiority or Other; p = 0.0383, Wilcoxon (Mann-Whitney)
Statistical Analysis 4: Comparison: Desoximetasone 0.25% Twice Daily vs Vehicle Twice Daily; Test type: Superiority or Other; p = 0.0154, Wilcoxon (Mann-Whitney)
Statistical Analysis 5: Comparison: Desoximetasone 0.05% Once Daily vs Desoximetasone 0.25% Once Daily; Test type: Superiority or Other; p = 0.1892, Wilcoxon (Mann-Whitney)
Statistical Analysis 6: Comparison: Desoximetasone 0.05% Twice Daily vs Desoximetasone 0.25% Twice Daily; Test type: Superiority or Other; p = 0.0010, Wilcoxon (Mann-Whitney)
Statistical Analysis 7: Comparison: Desoximetasone 0.05% Once Daily vs Desoximetasone 0.05% Twice Daily; Test type: Superiority or Other; p = 0.0363, Wilcoxon (Mann-Whitney)
Statistical Analysis 8: Comparison: Desoximetasone 0.25% Once Daily vs Desoximetasone 0.25% Twice Daily; Test type: Superiority or Other; p = 0.2162, Wilcoxon (Mann-Whitney)

ADVERSE EVENTS:
Time Frame: 6 months
Arm/Group | Desoximetasone 0.05% Once Daily | Desoximetasone 0.05% Twice Daily | Desoximetasone 0.25% Once Daily | Desoximetasone 0.25% Twice Daily | Vehicle Once Daily | Vehicle Twice Daily
Serious Adverse Events (participants affected / at risk) | 0/30 | 0/31 | 0/30 | 0/29 | 0/15 | 0/15
Other Adverse Events (participants affected / at risk) | 6/30 | 2/31 | 7/30 | 4/29 | 5/15 | 6/15
OTHER ADVERSE EVENTS (reported when occurring in more than 3% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Desoximetasone 0.05% Once Daily (N=30) | Desoximetasone 0.05% Twice Daily (N=31) | Desoximetasone 0.25% Once Daily (N=30) | Desoximetasone 0.25% Twice Daily (N=29) | Vehicle Once Daily (N=15) | Vehicle Twice Daily (N=15)
Application Site Dryness (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 2 (2) | 0 (0) | 2 (3) | 1 (2)
Application Site Erythema (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Application Site Irritation (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Application Site Pruritus (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Back Pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Excoriation (Skin and subcutaneous tissue disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Folliculitis (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Furuncle (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0) | 0 (0) | 0 (0)
Gastritis (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Headache (General disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0) | 0 (0) | 2 (2)
Hypercholesterolaemia (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Hypertension (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0)
Nasopharyngitis (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Nausea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Rash (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Tooth Infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Tooth Injury (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Tooth Ache (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Upper Respiratory Tract Infection (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No